CLINICAL TRIAL: NCT00893243
Title: Efficacy Comparative Study Between Tears Again®, o Opticol® e o Optive® in Clinical and Symptomatology Treatment of Dry Eye Syndrome in Contact Lens Wearers and/or Computers Users
Brief Title: Efficacy Comparative Study Between Tears Again®, Opticol® and Optive®
Status: Completed | Type: Observational
Sponsor: Hospital de Sao Sebastiao (Other)
Responsible Party: Dr Lilianne Duarte, MD, Ophthalmologist
Other Study IDs: HSS-01-08
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1Tears Again/Control
- 2Opticol/Control
- 3Optive/Control
- 4Tears Again/Opticol
- 5Tears Again/Optive
- 6Opticol/Optive

SUMMARY:
Primary Purpose:

* To compare the efficacy in treating dry eye syndrome in contact lens wearers or computer users of Tears Again® versus Opticol® versus Optive®

Secondary Purpose:

* Subjective evaluation of symptomatology
* Evaluation of preference in different kind of administration - spray versus monodoses versus multi-doses

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed
* Age >18 years and < 55 years
* Daily wearer of soft contact lens and/or daily (> 4 hours/day) computer user

Exclusion Criteria:

* Dry eye Syndrome other than of evaporative etiology, according to DEWS
* Ocular or systemic disease that can affect the normal tear film
* Pregnancy or pregnancy risk (no contraceptive method), lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Administrative staff of the hospital with more than 4 hours/day computer use and contact lens wearers
Sampling Method: Probability Sample
Enrollment: 27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilianne Duarte, MD, Principal Investigator — Ophthalmologist; José Salgado-Borges, PhD, Study Director — Ophthalmology Department Director
Locations (1):
- Serviço de Oftalmologia, Hospital de São Sebastião, Santa Maria da Feira, Portugal